CLINICAL TRIAL: NCT05435001
Title: Evolution of a New Algorithm of Heart Rate Variability Analysis From Two-channel Holter Electrocardiogram in Pre-diagnosis of Obstructive Sleep Apnea Syndrome: a Study on Diagnostic Accuracy
Brief Title: Screening of Sleep Apnea by Holter Electrocardiography: Validation of Heart Rate Variability Analysis Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Collaborators: Amatis Software and Fysiologic Smart ECG Solutions (Unknown)
Responsible Party: Principal Investigator, Zeynep Zeren Ucar, Professor Doctor, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGHCEAH-KAEK-139-2022730-35
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea Syndromes
Keywords: Heart rate variability, Holter ECG monitoring
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OSAS disease status (Experimental): The dependent variable was diseased status (OSAS +/-). The independent variables analyzed were age, sex, body mass index (BMI), and for HRV variables, their day and night values and the differences between their night and day values (D[D/N]), as night mean HR, D[D/N] mean HR, night r-MSSD, D[D/N] r-MSSD, night SDNN, D[D/N] SDNN, night SDNN index, D[D/N] SDNN index, night SDANN, and D[D/N] SDANN.
  Interventions: Device: Holter ECG Monitoring

INTERVENTIONS:
Device: Holter ECG Monitoring — Holter electrocardiogram monitoring will be carried out for 24 h simultaneously with the PSG monitoring using a 2- lead ambulatory electrocardiograph (Fysiologic; kind courtesy: MedTech Company, Amsterdam, Holland). We will calculate the time-domain, frequency-domain and non-linear indices by HRV. Several parameters describing the differences between RR intervals will be calculated: the square root of the mean of the sum of the squares of differences between adjacent normal RR intervals (r-MSSD), SD of NN intervals (SDNN), SD of the averages of NN intervals in all 5-minute segments of the recording (SDANN), and mean of the SD of all NN intervals for all consecutive 5-minute segments of the recording (SDNN index). All variables will be calculated for the 24-hour, daytime (2:00 to 9:00 PM), and nighttime (midnight to 7 AM) periods, and the differences between daytime and nighttime values (D[D/N]) will be computed.

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a growing health concern affecting up to 60 % of population with cardiovascular disease. Despite the high cardiovascular morbidity and mortality associated with this syndrome, the substantial inconvenience and cost of polysomnography recordings may delay routine evaluation. Polysomnography (PSG) is the gold standard for diagnosis. However, this is a costly and time-consuming examination. Sympathoadrenergic balance obtained from the routine Holter monitoring suggesting the presence of OSAS, can enable patients to be guided and their PSGs to be primarily held.Abnormalities in nocturnal cyclical heart rate (HR) variations have previously been described in sleep-related breathing disorders. Compared with PSG, holter electrocardiogram has the advantages of pervasion, lower cost, no need for overnight hospitalization, greater similarity to normal conditions, and good compliance. The observation of changes in heart rate associated with apneic events has a potential to be used as an alternative technique for identification of subjects with OSAS. In regard to the feasibility of screening OSAS by HRV analysis by holter electrocardiogram monitoring, it has already been reported that a 24-h electrocardiographic monitoring might be useful to diagnose OSAS. It became a more feasible technique to use following the development of a convenient recorder for OSAS screening by analyzing changes in heart rate.

DETAILED DESCRIPTION:
To find out whether a new algorithm of HRV analysis from holter ECG monitoring can be used as a screening test for the diagnosis of patients with moderate-to-severe risk of obstructive sleep apnea syndrome (OSAS) with an acceptable accuracy.For this, overnight sleep pattern will be investigated in at least 107 individuals by polysomnography and 24-h ambulatory electrocardiography. Heart rate variability sleep apnea risk score (HRV-SARS) will be calculated using HRV analyses.

The patients were recruited from individuals referred to our university hospital's sleep center for a polysomnography recording because of clinically suspected OSAS (with at least one of the following obstructive sleep apnea symptoms: witnessed apnea, snoring and/or daytime sleepiness) from May to July 2022. Prospectively 107 patients enrolled in the study according to inclusion and exclusion criteria. Exclusion criteria were permanent or paroxysmal atrial fibrillation, permanent pacemaker, history of other sleep disorders, severe cardiopulmonary disease, severe diabetes mellitus, autonomic dysfunction or major physical or mental ailments. All patients underwent both a full polysomnography recording and ECG Holter monitoring.

This new algorithm of HRV analysis from holter ECG monitoring may represent an accurate and inexpensive screening tool in clinically suspected OSAS patients and may help focus resources on those at the highest risk.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be recruited from individuals referred to our university hospital's sleep center for a polysomnography recording because of clinically suspected OSAS (with at least one of the following obstructive sleep apnea symptoms: witnessed apnea, snoring and/or daytime sleepiness)

Exclusion Criteria:

* Permanent or paroxysmal atrial fibrillation, permanent pacemaker, severe cardiopulmonary disease, severe diabetes mellitus, autonomic dysfunction or major physical or mental ailments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 24 hour
  The variation in time intervals between heart beats. HRV analysis (in time, frequency and nonlinear domains) with 2-channel Holter ECG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Z Ucar, Prof Dr, Principal Investigator — Izmir Dr Suat Seren Chest Disease and Surgery Training and Research Hospital
Locations (1):
- Izmir Dr Suat Seren Chest Disease and Surgery Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No